CLINICAL TRIAL: NCT03102593
Title: A Randomized, Double-blind, Placebo-controlled, Phase II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of ARGX-113 in Patients With Primary Immune Thrombocytopenia
Brief Title: A Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of ARGX-113 in Patients With ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1603; 2016-003038-26 (EudraCT Number)
Record Dates: First submitted 2017-03-14; First posted 2017-04-06 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — efgartigimod alfa

STUDY DESIGN:
Intervention Model Description: Protocol designed to evaluate one or more interventions for treating a disease, syndrome or condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARGX-113 Dose A + SoC (Experimental): Patients will be randomized in a 1:1:1 ratio to ARGX-113 (Dose A or Dose B) or placebo
  Interventions: Drug: ARGX-113
- ARGX-113 Dose B +SoC (Experimental): Patients will be randomized in a 1:1:1 ratio to ARGX-113 (Dose A or Dose B) or placebo
  Interventions: Drug: ARGX-113
- Placebo + SoC (Placebo Comparator): Patients will be randomized in a 1:1:1 ratio to ARGX-113 (Dose A or Dose B) or placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ARGX-113 — ARGX-113 (Dose A or Dose B) or matching placebo will be administered IV weekly
  Arms: ARGX-113 Dose A + SoC; ARGX-113 Dose B +SoC
Other: Placebo — ARGX-113 (Dose A or Dose B) or matching placebo will be administered IV weekly
  Arms: Placebo + SoC

SUMMARY:
The purpose of the study is to determine safety, efficacy, tolerability and Pharmacokinetics of ARGX-113 in Patients with Primary Immune Thrombocytopenia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase II study in which approximately 36 patients will be randomized in a 1:1:1 ratio to receive either ARGX-113 Dose A, or ARGX-113 Dose B body weight or placebo in 4 infusions administered 1-week apart in addition to Standard-of-Care (SoC) treatment. Patients aged 18 to 85 years (inclusive) with confirmed primary immune thrombocytopenia (ITP) who have a platelet count ˂ 30 × 109/L and who are receiving oral corticosteroids and/or permitted oral immunosuppressants and/or Thrombopoietin receptor (TPO-R) agonist as SoC which must be maintained on a stable dose and frequency for at least 4 weeks prior to Screening.

The study will include a 2-week Screening, a 3-week Treatment period, and an 21-week follow-up (FU) period. The study is followed by an open label period where patients will be given the option to be treated with ARGX-113 Dose A in cycles of 4 weekly infusions with a minimum of 4 weeks apart. Patients may receive rescue therapy during the study at the discretion the investigator when deemed medically necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 to ≤ 85 years.
2. Must receive SoC treatment for ITP that has been stable in dose and frequency for at least 4 weeks prior to Screening. SoC may include oral corticosteroids and/or permitted oral immunosuppressants and/or TPO-R agonist.
3. Confirmed diagnosis of ITP with blood platelet counts < 30 × 109/L and who have not experienced major bleeding in the last 4 weeks prior to Screening.

Exclusion Criteria:

1. Use of anticoagulants, or any drug with antiplatelet effect within 3 weeks prior to Screening.
2. Patients who have received any blood support or transfusion within 4 weeks prior to Screening.
3. Use of Intravenous immunoglobulin G (IVIg) or anti-D immunoglobulin treatment within 4 weeks prior to screening.
4. Use of recombinant thrombopoietin at any time.
5. Use of rituximab within 6 months prior to Screening. Use of any anti-CD20 other than rituximab at any time is not permitted.
6. Use of immunosuppressants is not permitted within 4 weeks prior to Screening, with the exception of the following oral immunosuppressants: azathioprine, danazol, mycophenolate mofetil, mycophenolate sodium which must have been stable for at least 4 weeks prior to Screening.
7. Use of any other biological therapy or investigational drug than those previously indicated within 3 months or 5 half-lives of the drug (whichever is longer) prior to Screening.
8. Received vaccinations within 4 weeks prior to Screening or planned during the study.
9. At Screening, have clinically significant laboratory abnormalities
10. History of any thrombotic or embolic event within 12 months prior to Screening.
11. Known auto-immune disease other than ITP.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of serious adverse events (SAEs). | After the first administration of Investigational Medicinal Product day 1 to 30 days of a patient's last visit.
  Changes from Baseline in vital signs, electrocardiogram parameters (ECGs), physical examination abnormalities and clinical laboratory assessments.

SECONDARY OUTCOMES:
Frequency and proportion of patients with initial response | Over the study period (up to 13 weeks).
  Mean change from Baseline in platelet counts

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Newland, Study Chair — Barts Hospital, Cancer Centre in London
Locations (30):
- Austria (2):
  - Vienna, Vienna
  - Wien, Vienna
- Belgium (2):
  - Leuven, Leuven
  - Mont-Godinne, Namur
- Czechia (2):
  - Brno, Brno
  - Praha, Prague
- France (3):
  - Bordeaux, Bordeaux
  - Grenoble, Grenoble
  - Paris, Paris
- Germany (3):
  - Berlin, Berlin
  - Hanover, Hanover
  - Tubingen, Tübingen
- Hungary (6):
  - Budapest, Budapest
  - Debrecen, Debrecen
  - Gyula, Gyula
  - Kaposvar, Kaposvár
  - Nyiregyhaza, Nyíregyháza
  - Pecs, Pécs
- Poland (3):
  - Lublin, Lublin
  - Opole, Opole
  - Wroclaw, Wroclaw
- Spain (4):
  - A Coruna, A Coruña
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia
- Ukraine (4):
  - Dnipro, Dnipro
  - Ivano-Frankivsk, Ivano-Frankivsk
  - Nikolaev, Mykolayiv
  - Uzhgorod, Uzhhorod
- London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Newland AC, Sanchez-Gonzalez B, Rejto L, Egyed M, Romanyuk N, Godar M, Verschueren K, Gandini D, Ulrichts P, Beauchamp J, Dreier T, Ward ES, Michel M, Liebman HA, de Haard H, Leupin N, Kuter DJ. Phase 2 study of efgartigimod, a novel FcRn antagonist, in adult patients with primary immune thrombocytopenia. Am J Hematol. 2020 Feb;95(2):178-187. doi: 10.1002/ajh.25680. Epub 2019 Dec 10. PMID 31821591